CLINICAL TRIAL: NCT03499236
Title: RELIEVE-HF TRIAL: REducing Lung congestIon Symptoms Using the v-wavE Shunt in adVancEd Heart Failure
Brief Title: Reducing Lung CongestIon Symptoms in Advanced Heart Failure
Acronym: RELIEVE-HF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: V-Wave Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL7018
Record Dates: First submitted 2018-03-29; First posted 2018-04-17 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomized treatment versus control (1:1). Control patients will be allowed to cross-over at the completion of the blinded phase. A parallel roll-in arm will enroll up to 2 patients per site in an open-label study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the randomized cohort, participants, the clinical team, and research staff managing the patient after randomization will be blinded to study assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Treatment (Experimental): Treatment arm patients will undergo a diagnostic right heart catheterization and invasive echocardiography to determine study eligibility followed by transseptal catheterization and V-Wave Shunt implantation
  Interventions: Device: V-Wave Interatrial Shunt
- Control (Other): Control arm patients will undergo a diagnostic right heart catheterization and invasive echocardiography to determine study eligibility, but will not have transseptal catheterization or shunt implantation.
  Interventions: Other: Control
- Roll in (Experimental): Roll in arm patients will undergo a diagnostic right heart catheterization and invasive echocardiography to determine study eligibility followed by transseptal catheterization and V-Wave Shunt implantation
  Interventions: Device: V-Wave Interatrial Shunt

INTERVENTIONS:
Device: V-Wave Interatrial Shunt — The V-Wave Interatrial Shunt System, includes a permanent implant placed during a minimally invasive cardiac catheterization procedure using its dedicated Delivery Catheter. The device is implanted through the fossa ovalis and straddles the interatrial septum.
  Arms: Roll in; Treatment
Other: Control — Right heart catheterization, invasive echocardiography.
  Arms: Control

SUMMARY:
The objective of the RELIEVE-HF study is to provide reasonable assurance of safety and effectiveness of the V-Wave Interatrial Shunt System by improving meaningful clinical outcomes in patients with New York Heart Association (NYHA) functional Class II, Class III, or ambulatory Class IV heart failure (HF), irrespective of left ventricular ejection fraction, who at baseline are treated with guideline-directed drug and device therapies.

DETAILED DESCRIPTION:
This is a prospective, multi-center, 1:1 randomized, patient and observer blinded clinical study, with a Shunt Treatment arm and a non-implant Control arm. A total of approximately 500 patients will be randomized. Patients and all research staff managing the patients after randomization will be blinded during follow-up for a minimum of 12 months to a maximum of 24 months. Control patients will have the opportunity to receive a shunt after 24 months once unblinding occurs, if they provide consent, and continue to meet inclusion/exclusion criteria. All implanted patients will be followed for a total of 5 years from the time of the study device implantation.

ELIGIBILITY:
Main Inclusion Criteria:

* Both heart failure with reduced ejection fraction (HFrEF) and heart failure with preserved ejection fraction (HFpEF) patients
* NYHA Class II, Class III, or ambulatory Class IV HF
* Receiving guideline directed medical and device therapy (GDMT) for heart failure
* For NYHA Class III and ambulatory Class IV, at least one prior hospitalization for heart failure within the last year or elevated BNP level of at least 300 pg/ml or NT-proBNP level of at least 1,500 pg/ml. BNP/NT-ProBNP levels corrected for BMI
* For NYHA Class II, must have both hospitalization and elevated BNP levels as above specifications

Main Exclusion Criteria:

* Systolic blood pressure <90 or >160 mmHg
* Presence of Intracardiac thrombus
* Pulmonary hypertension with PASP of ≥70 mm/Hg or PVR > 4 WU
* Significant RV dysfunction - TAPSE <12mm or RVFAC ≤25%
* Left Ventricular End-Diastolic Diameter (LVEDD) >8cm
* Moderate to severe aortic or mitral stenosis
* Stroke or TIA or DVT within the last 6 months
* eGFR <25 ml/min/1.73 m^2
* Anatomical anomaly on TEE or ICE that precludes implantation of Shunt across fossa ovalis (FO) of the interatrial septum
* Inadequate vascular access for implantation of shunt, e.g. femoral venous access for transseptal catheterization and inferior vena cava (IVC) is not patent
* Hemodynamic heart rhythm, or respiratory instability at time of Final Exclusion Criteria

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety-Percentage of Treatment patients experiencing major device-related adverse events | 30-days after randomization
  Percentage of Treatment group patients experiencing any device-related Major Adverse Cardiovascular or Neurological Events (MACNE) during the first 30-days after randomization, compared to a pre-specified Performance Goal
Effectiveness-Hierarchical composite of death, heart transplant or left ventricular assist device (LVAD) implantation, HF hospitalizations, worsening HF events treated as an outpatient, and change in Kansas City Cardiomyopathy Questionnaire (KCCQ) | Follow-up duration at endpoint analysis ranges from a minimum of 12 to a maximum of 24 months
  Treatment and Control groups will be compared using the Finkelstein-Schoenfeld method

SECONDARY OUTCOMES:
6MWT changes | Baseline to 12 months
  6MWT changes
KCCQ changes | Baseline to 12 months
  KCCQ changes
KCCQ changes | Baseline through study completion, maximum of five years
  KCCQ changes
Time to all-cause death, LVAD/Transplant, or heart failure hospitalization | Baseline through study completion, maximum of five years
  Time to all-cause death, LVAD/Transplant, or heart failure hospitalization
Time to all-cause death or first heart failure hospitalization | Baseline through study completion, maximum of five years
  Time to all-cause death or first heart failure hospitalization
Cumulative heart failure hospitalizations | Baseline through study completion, maximum of five years
  Cumulative heart failure hospitalizations
Time to first heart failure hospitalization | Baseline through study completion, maximum of five years
  Time to first heart failure hospitalization
Modified Primary Effectiveness Endpoint including all-cause death, LVAD/Transplant, HF Hospitalizations, and worsening HF events treated as outpatient but without KCCQ | Baseline through study completion, maximum of five years
  Modified Primary Effectiveness Endpoint including all-cause death, LVAD/Transplant, HF Hospitalizations, and worsening HF events treated as outpatient but without KCCQ

CONTACTS AND LOCATIONS:
Overall Officials: Stefan D Anker, MD, PhD, Principal Investigator — University Medical Center Gottingen, Germany; JoAnn Lindenfeld, MD, Principal Investigator — Vanderbilt University; Josep Rodés-Cabau, MD, Principal Investigator — Université Laval (CRIUCPQ-ULaval); Gregg W Stone, MD, Principal Investigator — Colombia University Medical Center
Locations (83):
- United States (43):
  - Abrazo Arizona Heart Hospital, Phoenix, Arizona
  - Arizona Heart Rhythm Center, Phoenix, Arizona
  - Scripps Health, La Jolla, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Keck Medical Center of USC, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Stanford Hospital, Stanford, California
  - Los Robles Hospital & Medical Center, Thousand Oaks, California
  - The Lundquist Institute (Harbor-UCLA) Medical Center, Torrance, California
  - South Denver Cardiology, Littleton, Colorado
  - Memorial Hospital, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - First Coast Cardiovascular Institute, Orange Park, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Midwest Cardiovascular Institute, Naperville, Illinois
  - St Elizabeth Medical Center, Edgewood, Kentucky
  - United Heart & Vascular Clinic, Saint Paul, Minnesota
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Valley Health System, Ridgewood, New Jersey
  - Weill Cornell, New York, New York
  - Rochester General Health System, Rochester, New York
  - Mission Hospital, Asheville, North Carolina
  - North Carolina Heart & Vascular, Raleigh, North Carolina
  - Summa Health, Akron, Ohio
  - Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Pinnacle / Pinnacle Health Cardiovascular Institute, Wormleysburg, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Centennial Medical Center, Nashville, Tennessee
  - Austin Heart, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - Texas Heart Institute, Houston, Texas
  - University of Texas Memorial Hermann, Houston, Texas
  - Methodist Hospital, San Antonio, Texas
  - Christus Mother Frances Hospital, Tyler, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Chippenham Medical Center, Richmond, Virginia
- Australia (4):
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Flinders Medical Centre, Adelaide
  - Prince Charles Hospital, Brisbane
  - St. Vincent's Hospital, Melbourne
- Belgium (2):
  - Ziekenhuis Aan De Stroom vzw (ZAS), Antwerp
  - AZ Sint-Jan Brugge, Bruges
- Canada (2):
  - Montréal Heart Institute, Montreal
  - Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec
- Germany (9):
  - Charité - Universitätsmedizin Berlin Campus Virchow-Klinikum, Berlin
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Vivantes Klinikum Urban, Berlin
  - Marienkrankrankenhas, Hamburg
  - Universitätsklinikum Leipzig, Leipzig
  - Herzzentrum Leipzig, Leipzig
  - Ludwig-Maximilians-Universität München, München
  - SANA Remscheid, Remscheid
  - University of Rostock, Rostock
- Israel (7):
  - University Hospital Samson Assuta Ashdod, Ashdod
  - Yitzhak Shamir Medical Center, Be’er Ya‘aqov
  - Hadassah Medical Center, Jerusalem
  - The Chaim Sheba Medical Center Tel-Hashomer, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - The Baruch Padeh Medical Center, Poriya, Tiberias
- Netherlands (3):
  - St Antonius Ziekenhuis Nieuwegein, Nieuwegein, Utrecht
  - Academic Medical Center, The Netherlands, Amsterdam
  - Erasmus University Medical Center Rotterdam, Rotterdam
- Christchurch Hospital, Christchurch, New Zealand
- Poland (3):
  - Institute of Cardiology, Warsaw, Warsaw
  - The 4th Military Clinical Hospital Wroclaw, Wroclaw
  - University Hospital Wroclaw, Wroclaw
- Spain (7):
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Badalona Barcelona, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Puerta de Hierro-Majadahonda, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
- Switzerland (2):
  - Bern University Hospital, Bern
  - University Hospital of Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zile MR, Abraham WT, Lindenfeld J, Anker SD, Rodes-Cabau J, Pfeiffer MP, Boehmer JP, Litwin S, Baicu CF, Villota JN, Lee EC, Holcomb R, O'Keefe P, Eigler NL, Stone GW; RELIEVE-HF Investigators. Mechanistic Basis for Differential Effects of Interatrial Shunt Treatment in HFrEF vs HFpEF: The RELIEVE-HF Trial. JACC Cardiovasc Imaging. 2026 Jan;19(1):1-15. doi: 10.1016/j.jcmg.2025.08.005. Epub 2025 Sep 15. PMID 40892630
- [Derived] Stone GW, Lindenfeld J, Rodes-Cabau J, Anker SD, Zile MR, Kar S, Holcomb R, Pfeiffer MP, Bayes-Genis A, Bax JJ, Bank AJ, Costanzo MR, Verheye S, Roguin A, Filippatos G, Nunez J, Lee EC, Laufer-Perl M, Moravsky G, Litwin SE, Prihadi E, Gada H, Chung ES, Price MJ, Thohan V, Schewel D, Kumar S, Kische S, Shah KS, Donovan DJ, Zhang Y, Eigler NL, Abraham WT; RELIEVE-HF Investigators. Interatrial Shunt Treatment for Heart Failure: The Randomized RELIEVE-HF Trial. Circulation. 2024 Dec 10;150(24):1931-1943. doi: 10.1161/CIRCULATIONAHA.124.070870. Epub 2024 Sep 23. PMID 39308371